CLINICAL TRIAL: NCT00477464
Title: Clinical Evaluation of Lapatinib Administered With Capecitabine in Japanese Patients With ErbB2 Overexpressing Advanced or Metastatic Breast Cancer
Brief Title: Lapatinib in Combination With Capecitabine in Japanese Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109749
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2011-09

CONDITIONS: Metastatic Breast Cancer; Neoplasms, Breast
Keywords: dual kinase inhibitor,; EGFR/ErbB1,; ErbB2-overexpressing,; GW572016,; advanced/metastatic breast cancer, Lapatinib,; HER-2/new,; pharmacokinetics
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib+capecitabine (Experimental): Lapatinib 1250mg once daily +capecitabine 2000mg/m^2 twice daily (14 days out of 21 days)
  Interventions: Drug: Lapatinib; Drug: capecitabine

INTERVENTIONS:
Drug: Lapatinib — 1250mg once daily
Drug: capecitabine — 2000mg/m^2 twice daily (14 days out of 21 days)

SUMMARY:
This study is to evaluate the safety and efficacy of lapatinib taken together with capecitabine in Japanese patients. The study will proceed in two phases; the first phase(Part1) will lead to an evaluation of the mainly tolerability as well as PK parameters. If there are no major safety concerns in Part 1, the study will move into the second phase (Part 2) to further evaluate the safety and clinical activity.

ELIGIBILITY:
Inclusion criteria:

* Subjects eligible for enrolment in the study must meet all of the following criteria:
* Patients who have consent to this study participation and signed into Informed consent form.
* Subjects must have histologically confirmed invasive breast cancer with stage IIIB, stage IIIC with T4 lesion, or stage IV disease.
* Documentation of ErbB2 overexpression [IHC3+ or IHC2+ with FISH confirmation] is required based on local laboratory.
* Subjects must have documented progressive advanced or metastatic breast cancer.
* Subjects must have refractory breast cancer defined as progression in the locally advanced or metastatic setting or relapse within 6 months of completing adjuvant therapy. Prior therapies must include, but are not limited to:
* Taxane containing regimen for at least 4 cycles or 2 cycles provided disease progression occurred while on taxane.
* Anthracycline containing regimen for at least 4 cycles or 2 cycles provided disease progression occurred while on anthracycline.
* Subjects who relapse >6 months after completion of adjuvant anthracycline-containing chemotherapy, and for whom further anthracycline is not indicated, will be considered to have met the anthracycline prior exposure requirement.
* Taxanes and anthracyclines may have been administered concurrently or separately.
* Prior treatment with capecitabine is not permitted.
* Prior treatment must have contained trastuzumab alone or in combination with other chemotherapy for at least 6 weeks of standard doses in the adjuvant or advanced/metastatic setting.
* Subjects with hormone receptor positive tumors must have disease progression following hormonal therapy unless intolerant to hormonal therapy or hormonal therapy is not considered to be clinically appropriate.
* Subjects with stable CNS metastases (asymptomatic, and off systemic steroids and anticonvulsants for at least 3 months) are eligible.
* Measurable disease according to modified RECIST (Response Evaluation Criteria in Solid Tumors) (see Section 6.2, Efficacy p.49).
* Subjects must have archived tumor tissue available for biomarker assessment.
* Female subjects must be ≥20
* ECOG Performance Status of 0 or 1.
* Life expectancy of ≥12 weeks.
* Measurable lesions may be in the field of prior irradiation. However, there must be at least a 4-week period between the last radiation treatment and the baseline scan documenting disease status for the lesion to be measurable.
* Cardiac ejection fraction within the institutional range of normal as measured by ECHO (or MUGA if ECHO is not available). If no institutional range is available, cardiac ejection fraction must be ≥50%.
* Adequate hematologic value, hepatic and renal function as defined below. Hematologic ANC (absolute neutrophil count) ≥1.5×109/L Hemoglobin ≥9 g/dL Platelets ≥100× 109/L Hepatic Serum bilirubin ≤1.5×ULN

  * 2.5×ULN if subject has Gilbert's syndrome AST and ALT ≤5×ULN if documented liver metastases
  * 3×ULN without liver metastases Renal Serum creatinine Creatinine clearance* ≤50 mL/min

    * Calculated by the Cockcroft and Gault Method

Exclusion criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Pregnant or lactating females.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. In addition, subjects with ulcerative colitis are excluded.
* History of other malignancy. Subjects who have been disease-free for at least 5 years or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior anticancer therapy.
* Active or uncontrolled infection.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Known history of uncontrolled or symptomatic angina, arrhythmia or congestive heart failure.
* No prior anti-ErbB1/ErbB2 inhibitor for breast cancer other than trastuzumab.
* Known history or clinical evidence of leptomeningeal carcinomatosis.
* Concurrent anticancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than capecitabine.
* Bisphosphonates for the treatment of bone metastases should not be initiated following the first dose of study medication. Prophylactic use of bisphosphonate in subjects without bone disease is not permitted, except for prevention of osteoporosis.
* Use of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication.
* Participation in other studies or use of other investigational drugs during this study.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to lapatinib or excipients of lapatinib.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to capecitabine, fluorouracil or any excipients.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Patients who an investigator judges ineligible to this study in consideration of patient's safety (e.g., complications).

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Japan (11):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib 1250 mg and Capecitabine 2000 mg/m^2: Participants took lapatinib and capecitabine. Lapatinib was orally administered at 1250 milligrams (mg) once daily. Capecitabine was orally administered at 1000 mg per square meter (mg/m^2) twice daily on the first day through the fourteenth day of each 21-day cycle.
Period: Overall Study
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Started | 51
Completed | 0
Not Completed | 51
Not completed — Lost to Follow-up | 1
Not completed — Death | 36
Not completed — Completion of protocol-defined follow-up | 14

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants] | 51

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Response (Independent Reviewer-assessed)
Description: CBR is defined as the percentage of participants receiving at least one dose of study medication who achieved a best overall response classified as a complete or partial (confirmed) tumor response or stable disease for at least 6 months (24 weeks). A "complete response" is defined as the disappearance of all target or non-target lesions, "partial response" and "disease progression" as at least a 30% decrease and at least a 20% increase, respectively, in the sum of the longest diameter of target lesions, and "stable disease" as neither "partial response" nor "disease progression."
Time Frame: Baseline, every 6 weeks until Week 24 and then every 12 weeks until disease progression (up to Week 119)
Population: Intent-to-treat (ITT) Population: participants who had received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 51
percentage of participants | 59
Statistical Analysis 1: Comparison: Lapatinib 1250 mg and Capecitabine 2000 mg/m^2; Test type: Superiority or Other; percentage of participants = 59, 95% CI 2-sided [44.2 to 72.4] — The estimated value represents the percentage of participants who achieved a best overall response of complete response, partial response, or stable disease

2. Secondary Outcome: Time to Progression (Independent Reviewer-assessed)
Description: Time to progression is defined as the interval between the start of treatment and the earliest date of disease progression or death due to breast cancer, if sooner. Time to progression was calculated by using the Kaplan Meier estimate.
Time Frame: Baseline, every 6 weeks until Week 24 and then every 12 weeks until disease progression or death due to breast cancer (up to Week 119)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Lapatinib 1250 mg and Capecitabine 2000 mg/m^2: Participants took lapatinib and capecitabine. Lapatinib was orally administered at 1250 mg once daily. Capecitabine was orally administered at 1000 mg/m^2 twice daily on the first day through the fourteenth day of each 21-day cycle.
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 51
weeks | 36.0 [27.1 to 48.0]

3. Secondary Outcome: Progression-free Survival (PFS) (Independent Reviewer-assessed)
Description: PFS is defined as the interval between the start of treatment and the earliest date of disease progression or death of any cause, if sooner.
Time Frame: Baseline, every 6 weeks until Week 24 and then every 12 weeks until disease progression or death (up to Week 119)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 51
weeks | 36.0 [27.1 to 48.0]

4. Secondary Outcome: 6-Month Progression-free Survival (Independent Reviewer-assessed)
Description: 6-Month progression-free survival is defined as the percentage of participants surviving without progressive disease at 6 months (24 weeks) after the start of treatment. Progressive disease is defined as at least a 20% increase in the sum of the longest diameter of target lesions.
Time Frame: Baseline and then every 6 weeks until Month 6 (Week 24)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 51
percentage of participants | 68.2

5. Secondary Outcome: Objective Response (Independent Reviewer-assessed)
Description: Objective response is defined as the percentage of participants achieving a best overall response classified as a complete or partial (confirmed) tumor response. Complete response is defined as the disappearance of all target or non-target lesions, and partial response is defined as at least a 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Baseline every 6 weeks until Week 24 and then every 12 weeks until disease progression or death (up to Week 119)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 51
percentage of participants | 24

6. Secondary Outcome: Overall Survival (Independent Reviewer-assessed)
Description: Overall survival is defined as the time from the start of treatment until death regardless of cause. For participants who did not die, time to death was censored at the time of last confirmation of survival.
Time Frame: Baseline and then followed every 4 weeks until death (up to Week 157.9) while on treatment. After treatment termination, followed every 12 weeks until death (up to Week 157.9)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 51
weeks | 78.6 [51.6 to 103.0]

7. Secondary Outcome: Time to Response (Independent Reviewer-assessed)
Description: Time to response is defined as the time from the start of treatment until the first documented evidence of complete response or partial response.
Time Frame: Baseline, every 6 weeks until Week 24 and then every 12 weeks until disease progression or death (up to Week 119)
Population: Participants in the ITT Population achieving a partial or complete response
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 12
weeks | 6.9 [5.4 to 11.6]

8. Secondary Outcome: Duration of Response (Independent Reviewer-assessed)
Description: For the subset of participants who showed a complete or partial response, duration of response is defined as the time from the first documented evidence of partial or complete tumor response until the first documented sign of disease progression or death due to breast cancer, if sooner.
Time Frame: Baseline, every 6 weeks until Week 24 and then every 12 weeks until disease progression or death (up to Week 119)
Population: Participants in the ITT Population achieving a partial or complete response
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 12
weeks | 42.7 [26.9 to 68.4]

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lapatinib
Description: Pharmacokinetic (PK) samples were collected at pre-dose, and at 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, 10, 12, and 24 hours (hr) (plus or minus 30 minutes) after dosing. Cmax is defined as the maximum concentration of lapatinib.
Time Frame: Week 2
Population: PK Population: consisted of the first six participants who were enrolled into the study and evaluable for the PK parameters of the investigational products. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms/milliliter (ng/ml)
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
nanograms/milliliter (ng/ml) | 3520.872 [2570.460 to 4822.694]

10. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Lapatinib
Description: PK samples were collected at pre-dose, and at 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, 10, 12, and 24 hr (plus or minus 30 minutes) after dosing. Tmax is defined as the time to peak concentration from initiation of lapatinib dosing.
Time Frame: Week 2
Population: PK Population. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
hr | 4.727 [3.264 to 6.847]

11. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Lapatinib
Description: Terminal elimination half-life is defined as the duration until observation of half of the maximum concentration. PK samples were collected at pre-dose, and at 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, 10, 12, and 24 hr (plus or minus 30 minutes) after dosing.
Time Frame: Week 2
Population: PK Population. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
hr | 11.948 [9.267 to 15.405]

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve Within the Dosing Interval AUC0-tau of Lapatinib
Description: PK samples were collected at pre-dose, and at 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, 10, 12, and 24 hr (plus or minus 30 minutes) after dosing. AUC is defined as the area under the concentration-time curve from 0 to last quantifiable concentration (AUC 0-tau). AUC is a measure of exposure.
Time Frame: Week 2
Population: PK Population. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/ml
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
hr*ng/ml | 48153.776 [34575.918 to 67063.618]

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to 24 Hours AUC0-24 of Lapatinib
Description: PK samples were collected at pre-dose, and at 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, 10, 12, and 24 hr (plus or minus 30 minutes) after dosing. AUC is defined as the area under the concentration-time curve from 0 to 24 hour after dosing (AUC 0-24). AUC is a measure of exposure.
Time Frame: Week 2
Population: PK Population. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/ml
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
hr*ng/ml | 48063.990 [34431.610 to 67093.788]

14. Secondary Outcome: Cmax of Capecitabine, 5'-Fluorouracil (5-FU), and Alpha-fluoro-beta-alanine (FBAL)
Description: PK samples were collected at pre-dose, and at 0.5 (plus or minus 5 minutes), 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, and 10 hr (plus or minus 30 minutes) after dosing. Cmax is defined as the maximum concentration of drug. 5-FU and FBAL were evaluated because of the following reasons: (1) capecitabine is an orally administered fluoropyrimidine carbamate selectively activated to fluorouracil (5-FU) in tumors; (2) FBAL is an inactive major metabolite of capecitabine, and metabolites of capecitabine are excreted mainly in urine.
Time Frame: Week 2
Population: PK Population. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
ng/ml
  Capecitabine | 2698.033 [1491.563 to 4880.371]
  5-FU | 282.967 [127.386 to 628.562]
  FBAL | 5771.578 [4999.139 to 6663.370]

15. Secondary Outcome: Tmax of Capecitabine, 5'-Fluorouracil (5-FU), and Alpha-fluoro-beta-alanine (FBAL)
Description: PK samples were collected at pre-dose, and at 0.5 (plus or minus 5 minutes), 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, and 10 hr (plus or minus 30 minutes) after dosing. Tmax is defined as the time to peak concentration from initiation of dosing. 5-FU and FBAL were evaluated because of the following reasons: (1) capecitabine is an orally administered fluoropyrimidine carbamate selectively activated to fluorouracil (5-FU) in tumors; (2) FBAL is an inactive major metabolite of capecitabine, and metabolites of capecitabine are excreted mainly in urine.
Time Frame: Week 2
Population: PK Population. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
hr
  Capecitabine | 1.305 [0.480 to 3.544]
  5-FU | 1.305 [0.480 to 3.544]
  FBAL | 2.899 [1.862 to 4.514]

16. Secondary Outcome: t1/2 of Capecitabine, 5'-Fluorouracil (5-FU), and Alpha-fluoro-beta-alanine (FBAL)
Description: Terminal elimination half-life is defined as the duration until observation of half of the maximum concentration. PK samples were collected at pre-dose, and at 0.5 (plus or minus 5 minutes), 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, and 10 hr (plus or minus 30 minutes) after dosing. 5-FU and FBAL were evaluated because of the following reasons: (1) capecitabine is an orally administered fluoropyrimidine carbamate selectively activated to fluorouracil (5-FU) in tumors; (2) FBAL is an inactive major metabolite of capecitabine, and metabolites of capecitabine are excreted mainly in urine.
Time Frame: Week 2
Population: PK Population. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
hr
  Capecitabine | 0.865 [0.438 to 1.709]
  5-FU | 0.838 [0.572 to 1.229]
  FBAL | 2.437 [2.100 to 2.828]

17. Secondary Outcome: AUC0-tau of Capecitabine, 5'-Fluorouracil (5-FU), and Alpha-fluoro-beta-alanine (FBAL)
Description: PK samples were collected at pre-dose, and at 0.5 (plus or minus 5 minutes), 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, and 10 hr (plus or minus 30 minutes) after dosing. AUC is defined as the area under the concentration-time curve from 0 to last quantifiable concentration (AUC 0-tau). 5-FU and FBAL were evaluated because of the following reasons: (1) capecitabine is an orally administered fluoropyrimidine carbamate selectively activated to fluorouracil (5-FU) in tumors; (2) FBAL is an inactive major metabolite of capecitabine, and metabolites of capecitabine are excreted mainly in urine.
Time Frame: Week 2
Population: PK Population. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/ml
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
hr*ng/ml
  Capecitabine | 3997.313 [3008.973 to 5310.288]
  5-FU | 514.670 [349.554 to 757.782]
  FBAL | 29035.744 [26354.157 to 31990.189]

18. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to 12 Hours (AUC0-12) of Capecitabine, 5'-Fluorouracil (5-FU), and Alpha-fluoro-beta-alanine (FBAL)
Description: PK samples were collected at pre-dose, and at 0.5 (plus or minus 5 minutes), 1, 2, 3, 4 (plus or minus 15 minutes), 6, 8, and 10 hr (plus or minus 30 minutes) after dosing. AUC is defined as the area under the concentration-time curve from 0 to 12 hours after dosing (AUC 0-12). 5-FU and FBAL were evaluated because of the following reasons: (1) capecitabine is an orally administered fluoropyrimidine carbamate selectively activated to fluorouracil (5-FU) in tumors; (2) FBAL is an inactive major metabolite of capecitabine, and metabolites of capecitabine are excreted mainly in urine.
Time Frame: Week 2
Population: PK Population. One participant was excluded due to dose reduction.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/ml
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 5
hr*ng/ml
  Capecitabine | 3999.383 [3011.222 to 5311.818]
  5-FU | 544.318 [366.956 to 807.405]
  FBAL | 30478.416 [27682.239 to 33557.034]

19. Secondary Outcome: Trough Concentration of Lapatinib
Description: PK samples were collected at pre-dose on Day 14 and Day 21 (minus 2 days). Trough concentration is defined as the minimum serum concentration at steady state after a repeated dose of lapatinib.
Time Frame: Week 2
Population: ITT Population. Evaluable samples were not taken from some participants.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 42
ng/ml
  Week 2, n=42 | 1065.558 (718.6293)
  Week 3, n=41 | 1243.540 (849.3387)

20. Secondary Outcome: Trough Concentration of Capecitabine, 5-FU, and FBAL
Description: PK samples were collected at pre-dose on Day 14 (minus 2 days). Trough concentration is defined as the minimum serum concentration at steady state after a repeated dose. 5-FU and FBAL were evaluated because of the following reasons: (1) capecitabine is an orally administered fluoropyrimidine carbamate selectively activated to fluorouracil (5-FU) in tumors; (2) FBAL is an inactive major metabolite of capecitabine, and metabolites of capecitabine are excreted mainly in urine.
Time Frame: Week 2
Population: ITT Population. Evaluable samples were not taken from some participants.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Number analyzed (Participants) | 42
ng/ml
  Capecitabine | NA (NA) — A mean cannot be calculated because the concentration was below the quantification limit.
  5-FU | NA (NA) — A mean cannot be calculated because the concentration was below the quantification limit.
  FBAL | 668.73 (456.403)

ADVERSE EVENTS:
Arm/Group | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2
Serious Adverse Events (participants affected / at risk) | 8/51
Other Adverse Events (participants affected / at risk) | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2 (N=51)
Left ventricular dysfunction (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Syncope (Nervous system disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1250 mg and Capecitabine 2000 mg/m^2 (N=51)
Anaemia (Blood and lymphatic system disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 4
Cheilitis (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 34
Nausea (Gastrointestinal disorders) | 17
Stomach discomfort (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 17
Malaise (General disorders) | 6
Pyrexia (General disorders) | 9
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Cellulitis (Infections and infestations) | 3
Cystitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 15
Paronychia (Infections and infestations) | 14
Alanine aminotransferase increased (Investigations) | 15
Aspartate aminotransferase increased (Investigations) | 15
Blood albumin decreased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 16
Haematocrit decreased (Investigations) | 3
Haemoglobin decreased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 4
Red blood cell count decreased (Investigations) | 8
Weight decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 14
White blood cell count increased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 17
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 15
Eczema (Skin and subcutaneous tissue disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4
Ingrowing nail (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 39
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 17
Rash (Skin and subcutaneous tissue disorders) | 20
Skin exfoliation (Skin and subcutaneous tissue disorders) | 7
Flushing (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.